CLINICAL TRIAL: NCT00000907
Title: A Study of Discontinuing Maintenance Therapy in Subjects With Disseminated Mycobacterium Avium Complex (DMAC)
Brief Title: A Study to Examine the Effects of Stopping Preventive Therapy for Disseminated Mycobacterium Avium Complex (DMAC) in HIV-Positive Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 393; AACTG 393
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2003-06

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Immunity, Cellular; Antibiotics, Macrolide; Mycobacterium avium Complex; CD4 Lymphocyte Count; Disease Progression; Anti-HIV Agents
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Disease Progression

SUMMARY:
The purpose of this study is to evaluate the effects of stopping preventive therapy for DMAC in HIV-positive patients who (1) have been treated for DMAC for at least 12 months and are now free of any signs of DMAC for at least 16 weeks, and (2) have improved immune systems (CD4 cell counts greater than or equal to 100 cells/mm3) due to anti-HIV drug therapy.

DMAC is a serious and sometimes life-threatening infection that usually affects only HIV-positive patients with CD4 cell counts (cells of the immune system that fight infection) less than 50 cells/mm3. It is recommended that people who are likely to get DMAC be placed on preventive medications which help reduce the risk of infection. New anti-HIV combination drug therapies can increase CD4 cell counts and can reduce the level of HIV in the blood. When CD4 counts are increased, risk of DMAC infection is less. This study examines whether it is possible to stop preventive therapy for DMAC when CD4 counts are high without placing individuals at risk for getting DMAC again.

DETAILED DESCRIPTION:
A growing body of evidence suggests AIDS-related morbidity and mortality significantly decrease where potent antiretroviral therapies are used. HAART (highly active antiretroviral therapy) seems to significantly reduce the incidence of MAC. This study tests the validity of those observations.

Peripheral blood cultures and bone marrow (aspirate) samples from 50 eligible patients previously diagnosed with disseminated Mycobacterium avium complex (DMAC) are assessed for microbiologic sterilization of MAC at the time of study entry. If either bone marrow or blood cultures test positive for MAC, patients are discontinued from study. If cultures prove sterile, patients receive 6 weeks of treatment and then discontinue MAC therapy at Week 6 (entry into Step 2 of study). They are then monitored for clinical signs and symptoms of MAC recurrence and for the presence of mycobacteria in blood cultures. In cases of increased viral load during study, modification of antiretroviral therapy is allowed at the discretion of the patient's provider.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have 2 CD4 cell counts greater than or equal to 100 cells/mm3 within 60 days and 14 days prior to entry. Measurements must be taken at least 24 hours apart.
* Have been treated for DMAC with a drug regimen including at least 2 antimycobacterial drugs for at least 12 months, and have been free of symptoms for at least 16 weeks prior to study entry.
* Have been on anti-HIV therapy for at least 16 weeks and have been on stable anti-HIV therapy for at least 8 weeks prior to study entry.
* Are at least 13 years old (need consent of parent or guardian if under 18).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have any active infection (unless they have been on stable chronic suppressive therapy for at least 3 months).
* Are pregnant.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aberg, Study Chair; Judith Currier, Study Chair
Locations (24):
- United States (24):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Aberg, C. A study of discontinuing maintenance therapy in subjects with disseminated Mycobacterium avium complex. Program and abstracts of the 9th Conference on Retroviruses and Opportunistic Infections. 9th Conference on Retroviruses and Opportunistic Infections. 2002, February 24-28; Seattle Washington (abstract no634)
- [Background] Aberg JA, Williams PL, Liu T, Lederman HM, Hafner R, Torriani FJ, Lennox JL, Dube MP, MacGregor RR, Currier JS; AIDS Clinical Trial Group 393 Study Team. A study of discontinuing maintenance therapy in human immunodeficiency virus-infected subjects with disseminated Mycobacterium avium complex: AIDS Clinical Trial Group 393 Study Team. J Infect Dis. 2003 Apr 1;187(7):1046-52. doi: 10.1086/368413. Epub 2003 Mar 14. PMID 12660918